CLINICAL TRIAL: NCT05535933
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II/III Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of HMPL-523 in the Treatment of Warm Antibody Autoimmune Hemolytic Anemia
Brief Title: HMPL-523 (Sovleplenib) in the Treatment of Warm Antibody Autoimmune Hemolytic Anemia
Acronym: wAIHA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-523-00CH1
Record Dates: First submitted 2022-08-31; First posted 2022-09-10 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Warm Antibody Autoimmune Hemolytic Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HMPL-523 (Experimental): Phase II: Eligible subjects will receive 300 mg HMPL-523 treatment once daily for 8 weeks and at least 16 weeks open-label treatment.
  Phase III: Eligible subjects will receive 300 mg HMPL-523 treatment once daily for 24 weeks and enter open-label phase in the opinion of the Investigator.
  Interventions: Drug: HMPL-523(300mg PO QD)
- Placebo (Placebo Comparator): Phase II: Eligible subjects will receive 300 mg HMPL-523 treatment once daily for 8 weeks and at least 16 weeks open-label treatment.
  Phase III: Eligible subjects will receive 300 mg HMPL-523 treatment once daily for 24 weeks and enter open-label phase in the opinion of the Investigator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HMPL-523(300mg PO QD) — HMPL-523(300mg PO QD)
  Other Names: Sovleplenib
  Arms: HMPL-523
Drug: Placebo — Placebo(300mg PO QD)
  Arms: Placebo

SUMMARY:
Phase II Study: To evaluate the safety and preliminary efficacy of HMPL-523 in adult patients with wAIHA

Phase III Studies: Confirmation of Efficacy safety and of HMPL-523 in Adult Patients With wAIHA

DETAILED DESCRIPTION:
Phase II Study: the proportion of patients with overall Hb response by Week 24

Phase III study: the proportion of patients who achieve a durable response by Week 24

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent form (ICF);
2. Males or females aged 18 to 75 years;
3. Patients diagnosed with primary wAIHA or secondary wAIHA whose underlying diseases are stable;
4. Organs in good function.

Exclusion Criteria:

1. Patients with other types of AIHA other than wAIHA;
2. Patients with secondary wAIHA with unstable underlying disease;
3. Patients with drug-induced secondary wAIHA;
4. Patients with infections requiring systemic treatment;
5. Patients previously treated with Syk inhibitors (e.g., fostamatinib);
6. Patients with known allergy to the active ingredients or excipients of the study drug;
7. Patients with serious psychological or mental disorder;
8. Alcoholic or drug abuser;
9. Female patients who are pregnant and lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Phase II: overall Hb response rate | 24Weeks
  Phase II: Overall Hb response rate: the proportion of patients with overall Hb response by Week 24

SECONDARY OUTCOMES:
Phase III: Durable Hb response rate | 24Weeks
  Phase III: Durable Hb response rate: the proportion of patients who achieve a durable response by Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Fengkui Zhang, professor, Principal Investigator — offices director
Locations (5):
- China (5):
  - Guangdong Provincial People's Hospital, Lanzhou, Gansu
  - The First affiliated hospital of nanchang uiversity, Nanchang, Jiangxi
  - Bethune First Hospital Of Jilin University, Changchun, Jilin
  - Peking Union Medical College Hospital, Beijing
  - Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
The results of this study can be published in core journals or international scientific conferences, and the primary investigators who make significant contributions to the implementation and management of this study and the personnel who makes great contributions to the design, interpretation or analysis of this study (such as the staffs or consultants of the sponsor) can have their authorship attribution. The sponsor promises to provide the manuscript to the investigator for review before publication of any result of the study. Investigators have to obtain the approval of the sponsor before submitting academic articles or abstracts. The study personnel have the right to publish results of this study, however, the requirement of protecting confidential information must be met.
  The confidential information is the property of the sponsor only, cannot be disclosed to others without the written approval of the sponsor, and cannot be used for other purposes.
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] Zhao X, Sun J, Zhang Z, Chen M, Gong T, He G, Li Y, Liu H, Li F, Li X, Zhou H, Wang X, Hong M, Lei L, Yin H, Luo X, Li Y, Fan S, Guo X, Shi MM, Su W, Zhang L, Han B, Zhang F. Sovleplenib in patients with primary or secondary warm autoimmune haemolytic anaemia: results from phase 2 of a randomised, double-blind, placebo-controlled, phase 2/3 study. Lancet Haematol. 2025 Feb;12(2):e97-e108. doi: 10.1016/S2352-3026(24)00344-2. Epub 2025 Jan 9. PMID 39799953